CLINICAL TRIAL: NCT01873287
Title: Predicting Persistent Postconcussive Problems in Pediatrics: A Clinical Prediction Rule Derivation and Validation Study
Brief Title: Predicting Persistent Postconcussive Problems in Pediatrics (5P)
Acronym: 5P
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Roger Zemek, Pediatric Emergentologist, Division of Emergency Medicine, Children's Hospital of Eastern Ontario
Other Study IDs: CIHR-302955, CIHR-287347
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Concussions; PCS
Keywords: Concussions; Persistent post-concussion symptoms; PCS; Clinical Prediction Rule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Concussion, a mild traumatic injury common in children and adolescents, is a complex pathophysiological process affecting the brain. The lay press is inundated with reports of tragic consequences of concussion, and children are not immune.

Persistent postconcussive symptoms (PCS) is defined as the persistence of somatic, cognitive, physical, psychological or behavioural changes lasting more than one month following injury. PCS significantly impacts children and their family's quality of life through school absenteeism, depressed mood and loss of activities.

Validated, easy-to-use prognosticators do not exist for clinicians to identify children at highest risk for PCS. As a result,physicians cannot accurately inform children and parents whether they should expect longer symptoms, nor initiate pharmacotherapy or other management to reduce the occurrence or severity of PCS.

The investigators objective is to derive and validate a clinical prediction rule for the development of PCS in children and adolescents presenting to the emergency department (ED) following acute head injury. The investigators have three aims: (1) determine PCS incidence at one-month follow-up in children aged 5-17 who sustain a concussion; (2) derive a rule to predict PCS from variables present in the history and physical examination; and, (3) assess the accuracy, reliability and acceptability of the prediction rule in a subsequent cohort. Using a prospective, multicentre study at nine large Canadian pediatric EDs, the investigators will recruit the largest prospective epidemiological cohort of children with concussions in the literature.

This work will provide rigorous evidence to determine PCS incidence in children and its impact on quality of life. The results will enable clinicians to identify children at highest risk for PCS, optimize treatment and provide families with realistic anticipatory guidance. This study will also establish a strong and vital evidence base to advance concussion research.

DETAILED DESCRIPTION:
The full protocol has been published in BMJ Open (open access):

Zemek R, Osmond MH, Barrowman N for PERC Concussion Team. Predicting and preventing postconcussive problems in paediatrics (5P) study: protocol for a prospective multicentre clinical prediction rule derivation study in children with concussion. BMJ Open. 2013 Aug 1;3(8). pii:e003550. doi: 10.1136/bmjopen-2013-003550. PubMed PMID: 23906960. https://www.ncbi.nlm.nih.gov/pubmed/23906960

The primary outcome results have been published in JAMA (open access):

Zemek R, Barrowman N, Freedman SB, Gravel J, Gagnon I, McGahern C, Aglipay M, Sangha G, Boutis K, Beer D, Craig W, Burns E, Farion KJ, Mikrogianakis A, Barlow K, Dubrovsky AS, Meeuwisse W, Gioia G, Meehan WP 3rd, Beauchamp MH, Kamil Y, Grool AM, Hoshizaki B, Anderson P, Brooks BL, Yeates KO, Vassilyadi M, Klassen T, Keightley M, Richer L, DeMatteo C, Osmond MH; Pediatric Emergency Research Canada (PERC) Concussion Team. Clinical Risk Score for Persistent Postconcussion Symptoms among Children With Acute Concussion in the ED. JAMA. 2016 Mar 8;315(10):1014-25. doi: 10.1001/jama.2016.1203. PubMed PMID: 26954410. http://dx.doi.org/10.1001/jama.2016.1203

ELIGIBILITY:
Inclusion Criteria:

Subjects presenting to one of the study hospital EDs after sustaining a head injury will be eligible if they:

* are aged 5 to 17 years;
* have a concussion, defined by Zurich consensus statement;22
* suffered the initial injury in the previous 48 hours;
* are proficient in English or French.

Exclusion Criteria: Patients will be excluded if they present with traumatic head injuries with any of the following:

* GCS ≤13; any abnormality on standard neuroimaging studies, including any positive head CT findings (Note: neuroimaging is not required, but may be performed by the clinician if thought to be clinically indicated);
* neurosurgical operative intervention, intubation or PICU care required;
* multi-system injuries with treatment requiring admission to hospital, operating room or procedural sedation in the ED (Note: admission to hospital for observation or management of ongoing concussion symptoms is not an exclusion criteria);
* severe chronic neurological developmental delay resulting in communication difficulties;
* intoxication at the time of ED presentation as per clinician judgment;
* no clear history of trauma as primary event (e.g., seizure, syncope or migraine as primary event);
* previously enrolled in this same study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects presenting to one the nine participating Canadian pediatric hospitals (IWK Health Sciences Centre (NS), CHU Sainte-Justine (PQ), Montreal Children's Hospital (PQ), Children's Hospital of Eastern Ontario (ON), The Hospital for Sick Children (ON), Children's Hospital of Western Ontario (ON), Children's Hospital of Winnipeg (MB), Stollery Children's Hospital (AB) and Alberta Children's Hospital (AB)) EDs after sustaining a head injury.
Sampling Method: Non-Probability Sample
Enrollment: 3063 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Zemek, MD, Principal Investigator — CHEO
Locations (9):
- Canada (9):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - IWK Health Sciences Centre, Halifax, Nova Scotia
  - Alberta Children's Hospital, Calgary, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Engel J, van Ierssel JJ, Osmond MH, Tsampalieros A, Webster R, Zemek R. Return to the Emergency Department Within 3 Months Following Pediatric Acute Concussion. J Head Trauma Rehabil. 2023 Jul-Aug 01;38(4):319-328. doi: 10.1097/HTR.0000000000000852. Epub 2023 Feb 28. PMID 36854112
- [Derived] Gagnon I, Teel E, Gioia G, Aglipay M, Barrowman N, Sady M, Vaughan C, Zemek R; PEDIATRIC EMERGENCY RESEARCH CANADA (PERC) 5P TEAM. Parent-Child Agreement on Postconcussion Symptoms in the Acute Postinjury Period. Pediatrics. 2020 Jul;146(1):e20192317. doi: 10.1542/peds.2019-2317. Epub 2020 Jun 4. PMID 32499388
- [Derived] Teel EF, Zemek RL, Tang K, Gioia G, Vaughan C, Sady M, Gagnon IJ; Pediatric Emergency Research Canada (PERC) Concussion Team. The Stability of Retrospective Pre-injury Symptom Ratings Following Pediatric Concussion. Front Neurol. 2019 Jun 27;10:672. doi: 10.3389/fneur.2019.00672. eCollection 2019. PMID 31316452
- [Derived] Zemek R, Osmond MH, Barrowman N; Pediatric Emergency Research Canada (PERC) Concussion Team. Predicting and preventing postconcussive problems in paediatrics (5P) study: protocol for a prospective multicentre clinical prediction rule derivation study in children with concussion. BMJ Open. 2013 Aug 1;3(8):e003550. doi: 10.1136/bmjopen-2013-003550. PMID 23906960

RESULTS

PARTICIPANT FLOW:
Groups:
- Derivation Arm; Validation Arm: Inclusion criteria. Subjects presenting to one of the study hospital EDs after sustaining a head injury will be eligible if they: (1) are aged 5 to 17 years; (2) have a concussion, defined by Zurich consensus statement; (3) suffered the initial injury in the previous 48 hours; (4) are proficient in English or French.
  Exclusion criteria. Patients will be excluded if they present with traumatic head injuries with any of the following: GCS ≤13; any abnormality on standard neuroimaging studies,; neurosurgical operative intervention, intubation or PICU care required; multi-system injuries with treatment requiring admission to hospital, operating room or procedural sedation in the ED; severe chronic neurological developmental delay resulting in communication difficulties; intoxication at the time of ED presentation as per clinician judgment; no clear history of trauma as primary event (e.g., seizure, syncope or migraine as primary event); previously enrolled in this same study.
Period: Overall Study
Arm/Group | Derivation Arm | Validation Arm
Started | 2006 | 1057
Completed | 1701 | 883
Not Completed | 305 | 174

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Derivation Cohort | Validation Cohort | Total
Number analyzed (Participants) | 2006 | 1057 | 3063
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.8 [8.9 to 14.6] | 12.3 [9.6 to 14.8] | 12.0 [9.2 to 14.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 765 | 440 | 1205
  Male | 1241 | 617 | 1858
Region of Enrollment [Number; unit: participants]
  Canada | 2006 | 1057 | 3063

OUTCOME MEASURES:

1. Primary Outcome: Count of Children Who Have Persistent Post-concussive Symptoms (PCS) at One-month Follow-up.
Description: The primary outcome is the number of of children aged 5 - 17 years who have PCS at one-month follow-up. A PCS case is defined as an increase from pre-concussion baseline of three or more symptoms on the validated PCSI at one-month (consistent with the ICD-10 definition of PCS).
Time Frame: 1 month
Population: Completed 1-month followup.
Measure: Count of Participants; unit: Participants
Groups:
- PPCS in Derivation: August 2013 to September 2014
- PPCS in Validation: October 2014 to June 2015
Arm/Group | PPCS in Derivation | PPCS in Validation
Number analyzed (Participants) | 1701 | 883
Participants | 510 | 291

2. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL) Total Score at 4-weeks Post-injury
Description: The PedsQL™ is a reliable and valid measure of health-related quality of life in healthy children and adolescents and those with acute and/or chronic health conditions. Parent versions exist for children aged 2 to 18 years (in 4 age groups) and child versions for those aged 5 and over. The inventory covers four domains: physical, emotional, social and school. Items are calculated and transformed into an overall score with a range of 0 to 100 points, with more points indicating better quality of life. This secondary outcome measure will be used to determine the impact of PCS on quality of life on patients and families.
Time Frame: 1 month
Population: Completed PedsQL at 1-month post-concussion.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Participants With PPCS: The primary outcome measure, PPCS, was defined in keeping with the International Statistical Classification of Diseases and Related Health Problems, Tenth Revision (ICD-10) definition of postconcussion syndrome, which requires persistence beyond 4 weeks of at least 3 symptoms compared with state of being prior to the injury. In the study, an individual symptom was defined as a positive difference between the patient-reported current minus the perceived preinjury symptom rating on PCSI; both were completed 28 days after the injury.
- Participants Without PPCS: Less than 3 symptoms compared with state of being prior to the injury at 28 days. In the study, an individual symptom was defined as a positive difference between the patient-reported current minus the perceived preinjury symptom rating on PCSI; both were completed 28 days after the injury.
Arm/Group | Participants With PPCS | Participants Without PPCS
Number analyzed (Participants) | 510 | 1157
units on a scale | 70.0 [67.7 to 72.3] | 80.3 [78.1 to 82.6]

3. Secondary Outcome: Neuropsychological Evaluation
Description: A separate battery of neuropsychological assessment measures will be administered to those children who choose to participate in this arm of the study. This battery includes measures of intelligence, language, visual-spatial/motor functions, attention, memory/working memory, executive functioning, academic achievement, as well as behavioural/socioemotional functioning.
Time Frame: 1 month and 3 month
Population: Participants assessed at 4- and 12-weeks post-injury using direct, standardized measures of intellectual functioning, verbal memory, executive functioning, attention/working memory, processing speed and fine motor abilities.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Children With Neuropsychological Impairment: Incidence of neuropsychological impairment was determined using the Neuropsychological Impairment (NPI) rule (Beauchamp et al., 2015) and multiple hierarchical logistic and linear regressions were performed to assess the contribution of pre-morbid factors, acute symptoms, and acute cognitive testing to neuropsychological impairment and performance.
Arm/Group | Number of Children With Neuropsychological Impairment
Number analyzed (Participants) | 311
Participants | 32

ADVERSE EVENTS:
Groups:
- Participants: All enrolled participants.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/3063
Serious Adverse Events (participants affected / at risk) | 0/3063
Other Adverse Events (participants affected / at risk) | 0/3063

LIMITATIONS AND CAVEATS:
Selection bias (children presenting to ED as compared to general primary care) may limit generalizability.

There is no control group (e.g., orthopedic injury) to compare symptom scores. Socio-economic status and race data were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No